CLINICAL TRIAL: NCT04566614
Title: Preventing Viral Pandemic Associated Risk of Cancer Death Using Less Invasive Diagnostic Tests- Liquid Biopsies
Acronym: PREVAILctDNA
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 5292
Record Dates: First submitted 2020-06-02; First posted 2020-09-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Neoplasm, Colorectal; Neoplasm of Lung; Neoplasm, Bladder; Neoplasms Pancreatic; Biliary Tract Neoplasms; Gastro Intestinal Stromal Tumour
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- Biliary Tract Cohort: Patients with suspected biliary tract cancer will be offered ctDNA to support a diagnosis in patients with suspected early stage, locally advanced and advanced disease. This includes patients with tumours that are technically challenging to access with invasive biopsy or due to limitations in endoscopic ultrasound due to the COVID-19 pandemic. Patients with histological diagnosis will not be eligible for this study. Patients with suspected cancer will have ctDNA result (positive or negative) discussed at MDT in conjunction with PREVAIL-imaging risk stratification pathway to risk stratify in terms of cancer risk (low, intermediate and high risk), serum tumour markers and patient presentation which will dictate the appropriate treatment. Those with metastatic disease will have their treatment decision based on ctDNA result, radiology and patient characteristics after discussion between the treating clinician and patient
  Interventions: Other: ctDNA blood sampling
- Bladder Cancer Cohort: Patients with suspected bladder cancer (localised and metastatic) will be offered ctDNA to support their diagnosis, in cases where cystoscopy and biopsy are difficult to obtain due to the COVID-19 pandemic. Patients with histological diagnosis will not be eligible for this study. A positive ctDNA result will be supportive of a diagnosis of bladder cancer, their treatment may be prioritised and decided based on this result in conjunction with radiological findings, patient presentation and after discussion between the treating physician and patient
  Interventions: Other: ctDNA blood sampling
- Pancreatic Cancer Cohort: Patients with suspected pancreatic cancer will be offered ctDNA to support a diagnosis in patients with suspected early stage, locally advanced and advanced disease. This includes patients with tumours that are technically challenging to access with invasive biopsy or due to limitations in endoscopic ultrasound due to the COVID-19 pandemic. Patients with histological diagnosis will not be eligible for this study. Patients with suspected cancer will have ctDNA result (positive or negative) discussed at MDT in conjunction with PREVAIL-imaging risk stratification pathway to risk stratify in terms of cancer risk (low, intermediate and high risk), serum tumour markers and patient presentation which will dictate the appropriate treatment. Those with metastatic disease will have their treatment decision based on ctDNA result, radiology and patient characteristics after discussion between the treating clinician and patient
  Interventions: Other: ctDNA blood sampling
- Gastrointestinal Stromal Tumour Cohort: Those with suspected Gastrointestinal Stromal Tumour Cohort (GIST) are eligible for this study. KIT and PDGFR mutation detected using ctDNA in conjunction with radiological features will be supportive of a diagnosis of GIST. This may allow for the use of directed targeted therapy, or prioritise surgical resection in some cases. Patients with histological diagnosis will not be eligible for this study. However, patients with inadequate tissue for KIT/PDGFR analysis will be eligible for PREVAIL-ctDNA to confirm the diagnosis of GIST and help guide treatment decisions
  Interventions: Other: ctDNA blood sampling
- Lung Cancer Cohort: The use of ctDNA in the diagnosis and adaptive management of patients with lung cancer is well established, however not funded by NHS. As aerosol-generating bronchoscopy procedures have reduced due to the COVID-19 pandemic, patients with suspected lung cancer may be offered ctDNA to support the diagnosis. A positive ctDNA result in conjunction with radiological findings will assist in prioritising those suitable for upfront surgical resection, radiotherapy or systemic anti-cancer treatment. It may provide sufficient genotypic information to guide standard of care targeted therapies (usually two tests are required - biopsy and then next generation sequencing of extracted DNA), including in patients without sufficient tissue for EGFR and ALK testing which can be detected using ctDNA. The use of ctDNA to guide treatment decisions in this cohort will not require signed consent as it is considered a standard approach (not yet NHS funded)
  Interventions: Other: ctDNA blood sampling
- Colorectal Cancer Cohort: Patients with suspected colorectal cancer will often be referred following either suspicion on imaging or faecal immunochemical testing (FIT). FIT testing results will be used to prioritise patients for screening colonoscopy, in conjunction with the PREVAIL-imaging risk stratification pathway
  Interventions: Other: ctDNA blood sampling
- Part 2 Cohort: Patients with suspected advanced pancreatic or biliary tract cancer who have ctDNA via the ACCESS implementation pathway. The results must be deemed consistent with or diagnostic of pancreatic/biliary tract cancer by the molecular tumour board, discussed at central MDT and the patient cannot have a histological diagnosis.

INTERVENTIONS:
Other: ctDNA blood sampling — Screening/baseline blood sample to be analysed for ctDNA
  Groups: Biliary Tract Cohort; Bladder Cancer Cohort; Colorectal Cancer Cohort; Gastrointestinal Stromal Tumour Cohort; Lung Cancer Cohort; Pancreatic Cancer Cohort

SUMMARY:
The purpose of this study is to investigate the feasibility of using ctDNA to support cancer diagnosis and risk stratification where invasive aerosol generating testing (and/or tissue biopsy) is challenging due to infection risk, technical impracticalities and resource limitations, such as during the COVID-19 pandemic and the subsequent recovery period.

DETAILED DESCRIPTION:
This is a prospective, single-centre cohort pilot study using ctDNA informed treatment decisions. If the pilot study is successful within certain tumour types then this protocol may be extended to investigate further the benefit of ctDNA informed treatment decision in those tumour types.

Patients with suspected malignancy for whom invasive biopsy for definitive histological diagnosis is challenging either due to COVID-19-related resource limitations, infection control or technical feasibility will be considered for this study. In this setting liquid biopsy may be used in lieu of tissue biopsy to facilitate treatment or may be used to prioritise standard of care invasive diagnostic tests. The former includes patients who require repeat biopsies for genomic analysis following non-informative results where these would inform standard of care treatment (i.e. NICE (National Institute for Health and Care Excellence)/Cancer Drug Fund (CDF) approved drugs). Tumour types included in this study are therefore those where invasive aerosol generating diagnostic tests such as bronchoscopy, gastrointestinal endoscopy (including endoscopic ultrasound (EUS)) are part of the standard diagnostic pathway and where capacity for these tests has become severely constrained during (and likely after) the COVID-19 pandemic. Tumour types affected include some suspected biliary tract, bladder, colorectal, GIST, lung and pancreatic cancers.

The study is planned to continue until a total of 144 patients have been enrolled. This is anticipated to take up to 12-18 months. Follow-up will continue until patients have diagnosis made (based on ctDNA result) and treatment decision made (deferred or immediate).

Potential patients will be identified in and will usually at the multidisciplinary team (MDT) meeting. They will give consent to participate in the trial and offered a liquid biopsy (ctDNA) in lieu of a tissue biopsy if considered suitable for PREVAIL - ctDNA. This may include patients who require repeat biopsies for further genomic analyses when repeat biopsies are not feasible where liquid biopsy may support prioritisation for invasive diagnostics earlier. ctDNA analysis will involve copy number variant detection and low coverage whole genomic sequencing. ctDNA gene panels have already been validated against tissue based molecular diagnostics for paediatrics (ct_PAED) and colorectal cancer (ct_GI).

This analysis will be performed in an accredited clinical diagnostic laboratory (Translational Research Laboratory, Institute of Cancer Research). Patients will be stratified for treatment or further investigation based on their ctDNA result (either positive or negative), suspected tumour type, radiological (including PREVAIL-imaging risk stratification pathway) and clinical characteristics.

PREVAIL ctDNA- Part 2 Study:

PREVAIL part 2 is a multi-centre, prospective study assessing the impact of Guardant360© liquid biopsy in patients with radiologically suspicious pancreatic cancer (PC) and biliary tract cancer (BTC)without histological confirmation of malignancy.

Liquid biopsies will be implemented into the routine diagnostic pathway across 6 RMP sites for patients with radiologically suspicious stage III/IV PC/BTC as part of the ACCESS implementation programme. Over 12 months, approximately 650 patients will be identified at individual sites by the local team when seen for an invasive procedure and referred in parallel to the Guardant360© test. These patients will proceed through an invasive diagnostic pathway as is standard of care and have a liquid biopsy as a new standard of care. Most patients will undergo both invasive tissue biopsy and liquid biopsy.

Patients with informative liquid biopsy result, but without a histological diagnosis of cancer (either due to inconclusive biopsy result or if the invasive procedure hasn't been performed) will be considered suitable for the study. Only patients with detectable ctDNA without histological confirmation will be suitable for this study (approximately ¼ of patients entering the ACCESS programme). The study is planned to run parallel to the ACCESS implementation programme and it aims to enrole 150 patients.

As part of this study, treatment may be recommended based on the liquid biopsy result. Patients with an invasive biopsy result which is suitable to guide treatment will not be eligible.

ctDNA results will be discussed at the molecular tumour board (MTB) to provide clinical context and validity of the genomic result. In addition, all patients will be discussed at a central upper gastrointestinal cancer multidisciplinary team meeting (MDM) to discuss treatment based on ctDNA results. Treating clinicians will have access to the MTB outcome and patients may be treated based on the ctDNA result in the context of symptoms, tumour markers, and imaging results as a complete diagnostic package.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥18 years old
* Patients with suspected malignancies of early stage colorectal cancer (FIT intermediate and high risk), early and late stage pancreatic cancer, biliary tract cancer, gastro-intestinal stromal tumours, lung cancer or bladder cancer, without a definitive histological diagnosis (including those with inconclusive biopsy result) or
* Patients with histological diagnosis of lung cancer without adequate tissue for NHS genomic test directory predictive biomarker testing
* Ability to provide informed consent.
* Patients with performance status suitable for oncological treatments (ECOG performance status 0-2).

Exclusion criterion:

• Patients with an established histological diagnosis adequate to support standard of care treatment

PART 2:

Inclusion criteria

* Included in the ACCESS implementation programme
* Has detectable ctDNA on Guardant360© assay
* Discussion at molecular tumour board and central multi-disciplinary meeting confirming ctDNA variant is supportive of diagnosis of PC/BTC (diagnostic or consistent with)
* Performance status suitable for oncological treatment
* Ability to provide informed consent

Exclusion criteria

1. Previously diagnosed invasive or haematological malignancy within the past 3 years
2. Outcome at the molecular tumour board not supportive of cancer diagnosis (possibly consistent or not consistent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected malignancy for whom invasive biopsy for definitive histological diagnosis is challenging either due to COVID-19-related resource limitations, infection control or technical feasibility will be considered for this study
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
ctDNA detection rate within different cancer types (and overall) | Throughout study completion, up to one year
  The primary endpoint, ctDNA detection rate, overall and within different cancer types will be presented as a proportion of patients with a positive ctDNA test out of those tested, with 90% confidence intervals
PREVAIL ctDNA Part 2 Study | To run parallel for 12 months alongside the ACCESS implementation programme
  Primary end point, Proportion of patients with detectable ctDNA which supports a diagnosis of malignancy and commence treatment

SECONDARY OUTCOMES:
Proportion of patients with a positive ctDNA result which identified a diagnosis and/or commenced treatment | Throughout study completion, up to one year
  All secondary endpoints will be analysed in the patients diagnosed with suspected cancer, i.e. positive ctDNA result, unless stated. They will also be presented overall and by cancer type. The proportion of patients with positive ctDNA result which identified a diagnosis and/or commenced treatment will be presented as a proportion with 90% confidence intervals
Proportion of patients with a positive ctDNA result which assisted in prioritising invasive diagnostic tests | Throughout study completion, up to one year
  Proportion of patients with positive ctDNA result which assisted in prioritising invasive diagnostic tests will be presented as a proportion with 90% confidence intervals
The association of ctDNA result (positive versus negative) and the PREVAIL-imaging pathway scoring result | Throughout study completion, up to one year
  The association between ctDNA result (positive versus negative) and the PREVAIL-imaging pathway scoring result will be assessed descriptively by presenting cross-tabulations and relevant proportions
Estimation of the cost of liquid biopsy in lieu of tissue biopsy as compared to standard of care investigations and treatments prioritisation | Throughout study completion, up to one year
  Simple estimation of the cost of liquid biopsy in lieu of tissue biopsy as compared to standard of care investigations and treatments prioritisation will be performed
PREVAIL ctDNA Part 2 Study secondary end point 1a | To run parallel for 12 months alongside the ACCESS implementation programme
  Treatment response objective response rate
PREVAIL ctDNA Part 2 Study secondary end point 1b | To run parallel for 12 months alongside the ACCESS implementation programme
  Progression free survival
PREVAIL ctDNA Part 2 Study secondary end point 1c | To run parallel for 12 months alongside the ACCESS implementation programme
  Overall survival
PREVAIL ctDNA Part 2 Study secondary end point 2 | To run parallel for 12 months alongside the ACCESS implementation programme
  Proportion of patients who undergo a repeated invasive procedure
PREVAIL ctDNA Part 2 Study secondary end point 3a- comparison with NHS targets | To run parallel for 12 months alongside the ACCESS implementation programme
  Comparison of diagnostic pathway duration with NHS faster Diagnostic Standard (FDS)
PREVAIL ctDNA Part 2 Study secondary end point 3b- comparison with NHS targets | To run parallel for 12 months alongside the ACCESS implementation programme
  Comparison of diagnostic pathway duration with 62 day wait target
PREVAIL ctDNA Part 2 Study secondary end point 4a | To run parallel for 12 months alongside the ACCESS implementation programme
  Type of complications from invasive diagnostic procedures
PREVAIL ctDNA Part 2 Study secondary end point 4b | To run parallel for 12 months alongside the ACCESS implementation programme
  Frequency of complications from invasive diagnostic procedures
PREVAIL ctDNA Part 2 Study secondary end point 4c | To run parallel for 12 months alongside the ACCESS implementation programme
  Severity of complications from invasive diagnostic procedures
PREVAIL ctDNA Part 2 Study secondary end point 5 | To run parallel for 12 months alongside the ACCESS implementation programme
  Number and type of invasive procedures performed
PREVAIL ctDNA Part 2 Study secondary end point 5b | To run parallel for 12 months alongside the ACCESS implementation programme
  Number of histopathology reviews
PREVAIL ctDNA Part 2 Study secondary end point 5c | To run parallel for 12 months alongside the ACCESS implementation programme
  Number of tissue based NGS performed
PREVAIL ctDNA Part 2 Study secondary end point 6a | To run parallel for 12 months alongside the ACCESS implementation programme
  Healthcare costs associated with diagnostic pathway
PREVAIL ctDNA Part 2 Study secondary end point 6b | To run parallel for 12 months alongside the ACCESS implementation programme
  Cost per-quality adjusted-life-year of diagnostic pathway
PREVAIL ctDNA Part 2 Study secondary end point 6c | To run parallel for 12 months alongside the ACCESS implementation programme
  Number of hospital visits in diagnostic pathway
PREVAIL ctDNA Part 2 Study secondary end point 6d | To run parallel for 12 months alongside the ACCESS implementation programme
  Length of hospital stay during diagnostic pathway

CONTACTS AND LOCATIONS:
Overall Officials: Justin Mencel, MBBS, Principal Investigator — Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided